CLINICAL TRIAL: NCT02378441
Title: A Randomized, Open-labeled, Single-dose, Crossover Design Clinical Trial to Evaluate Pharmacokinetics and Safety of CJ-30056 20/750mg and Co-administration of Lipitor® 20mg and Glucophage SR 750mg in Fed Healthy Male Subjects
Brief Title: Phase 1 Study to Compare the Safety, Pharmacokinetic Profiles of CJ-30056 and Lipitor 20mg/Glucophage SR 750mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_ATM_105
Record Dates: First submitted 2015-02-16; First posted 2015-03-04 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Atorvastatin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ-30056 20/750mg (Experimental): fixed-dose combination of Atorvastatin 20mg and Metformin SR 750mg
  Interventions: Drug: Atorvastatin 20mg and Metformin SR 750mg; Drug: CJ-30056 20/750mg
- Atorvastatin 20mg and Metformin SR 750mg (Experimental): co-administration of Atorvastatin 20mg and Metformin SR 750mg
  Interventions: Drug: Atorvastatin 20mg and Metformin SR 750mg; Drug: CJ-30056 20/750mg

INTERVENTIONS:
Drug: Atorvastatin 20mg and Metformin SR 750mg — co-administration of Atorvastatin 20mg and Metformin SR 750mg
  Other Names: Atorvastatin (Lipitor) and Metformin (Glucophage SR)
Drug: CJ-30056 20/750mg — fixed-dosed combination of Atorvastatin 20mg and Metformin SR 750mg
  Other Names: not yet approved

SUMMARY:
This study is designed to evaluate safety and pharmacokinetic properties of the two treatments, the administration of CJ-30056 and the co-administration of atorvastatin 20mg and metformin SR 750mg, in healthy volunteers.

DETAILED DESCRIPTION:
To evaluate the bioequivalence of of CJ-30056 and co-administration of atorvastatin 20mg and metformin SR 750mg

ELIGIBILITY:
Inclusion Criteria:

1. Willing to adhere to protocol requirements and sign a informed consent form
2. Male volunteers in the age between 19 and 55 years old and have the weight range is not exceed ±20% of ideal weight
3. Subjects with no history of any significant chronic disease
4. Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data

Exclusion Criteria:

1. Use of barbital inducer or inhibitor medication within the 28 days before dosing
2. Symptom of an acute illness within 28 days prior to drug administration
3. History of clinically significant hepatic, renal, gastrointestinal diseases which might significantly interfere with ADME
4. History of surgery except or gastrointestinal diseases which might significantly change absorption of medicines
5. History of clinically significant allergies including drug allergies
6. History of clinically significant allergies about atorvastatin or metformin
7. Subjects who have ever or have plan to do intravenous injection of contrast medium (intravenous urography, intravenous cholangiography, computed tomography using contrast medium) within 28 days prior to drug administration
8. History of myopathy
9. Subjects who have genetic problems (galactose intolerance, Lapp lactase deficiency, glucose-galactase malabsorption etc.)
10. Clinical laboratory test values are outside the accepted normal range

    * AST or ALT >1.25 times to normal range
    * Total bilirubin >1.5 times to normal range
    * e-GFR <90 mL/min
11. History of drug, caffein(caffein > 400mg/day), smoking (cigarette > 10/day) or alcohol abuse(alcohol > 30 g/day)or Subjects who have ever drink within 7 days prior to drug administration
12. Special diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice) within 7 days prior to drug administration
13. Donated blood within 60 days prior to dosing
14. Participated in a previous clinical trial within 60 days prior to dosing
15. Use of any other medication, including herbal products, within 10 days before dosing
16. Subjects considered as unsuitable based on medical judgement by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of Atorvastatin and Metformin | Up to 32 hours

SECONDARY OUTCOMES:
Area under the curve(AUC) of Atorvastatin and Metformin | Up to 32 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jong-lyul Ghim, MD.PhD, Principal Investigator — Inje University Busanpaik Hospital

IPD SHARING:
Plan to Share IPD: No